CLINICAL TRIAL: NCT00371020
Title: The Effect of 5-FU and LMW Heparin on the Rate of Retinal Redetachment After Silicone Oil Removal in Cases of PVR
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Shahid Beheshti University of Medical Sciences (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 8373
Record Dates: First submitted 2006-08-31; First posted 2006-09-01 (Estimated); Last update posted 2007-07-12 (Estimated); Status verified 2007-07

CONDITIONS: Proliferative Vitreoretinopathy
Keywords: silicone oil; PVR; retinal redetachment; low molecular weight heparin; 5-FU
MeSH Terms: conditions — Vitreoretinopathy, Proliferative | interventions — Heparin, Low-Molecular-Weight; Fluorouracil

INTERVENTIONS:
Drug: low molecular weight heparin, 5-FU

SUMMARY:
To evaluate the effect of combined 5-FU and low molecular weight heparin in infusion on the rate of retinal redetachment after silicone oil removal in cases of proliferative vitreoretinopathy (PVR).

ELIGIBILITY:
Inclusion Criteria:

* Cases with history of vitrectomy and silicone oil injection for management of PVR who undergo silicone oil removal

Exclusion Criteria:

* any sign of retinal redetachment before silicone oil removal
* any sign of diabetic retinopathy

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2005-02; Study Completion 2007-07 (Estimated)

PRIMARY OUTCOMES:
Retinal redetachment rate

SECONDARY OUTCOMES:
visual acuity
intraocular pressure
reoperation
relative afferent pupillary defect

CONTACTS AND LOCATIONS:
Overall Officials: Hamid Ahmadieh, MD, Principal Investigator — Ophthalmic Research Center of Shaheed Beheshti Medical University
Locations (1):
- Hamid Ahmadieh, MD, Tehran, Tehran Province, Iran